CLINICAL TRIAL: NCT03386643
Title: Effect of the Probiotic Bifidobacterium Animalis Subsp. Lactis HN019 on Clinical, Histopathological and Immunophenotypic Features of Oral Lichen Planus
Brief Title: Effect of Bifidobacterium Animalis Subsp. Lactis HN019 on Oral Lichen Planus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ana Carolina Fragoso Motta, DDS, PhD, Teacher of Oral Diagnosis-Department of Stomatology, Public Oral Health and Forensic Dentistry, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAAE: 63003716.2.0000.5419
Record Dates: First submitted 2017-12-02; First posted 2017-12-29 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Oral Lichen Planus
Keywords: Oral lichen planus; Probiotics; Immunomodulation.
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Probiotics; Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: Symptomatic patients presenting OLP will be randomly assigned to either topical Bifidobacterium animalis subsp lactis HN019 or clobetasol propionate 0.05%, and they will receive capsules to be diluted in 15 ml of water containing 6 x 109 CFUs of Bifidobacterium subsp. lactis HN019 (experimental group) or 0.05% clobetasol propionate (control group) for mouth washing, twice a day for 4 weeks.
Who Masked: Participant, Investigator
Masking Description: Both patients and investigators who will assess the outcomes have no knowledge of the interventions assigned to individual participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bifidobacterium animalis subsp. lactis (Experimental): Intervention:
  Bifidobacterium animalis subsp. lactis HN019
  Interventions: Drug: Bifidobacterium animalis subsp. lactis HN019
- Clobetasol propionate 0.05% (Active Comparator): Intervention:
  Clobetasol propionate 0.05%
  Interventions: Drug: Clobetasol propionate 0.05%

INTERVENTIONS:
Drug: Bifidobacterium animalis subsp. lactis HN019 — The selected patients will receive capsules to be diluted in 15 ml of water containing 6 x 109 CFUs of Bifidobacterium subsp. lactis HN019 for mouthwash twice a day for 4 weeks.
  Other Names: Probiotic
  Arms: Bifidobacterium animalis subsp. lactis
Drug: Clobetasol propionate 0.05% — The selected patients will receive capsules to be diluted in 15ml of water containing clobetasol propionate 0.05% for mouthwash twice a day for 4 weeks.
  Other Names: Topical corticosteroid
  Arms: Clobetasol propionate 0.05%

SUMMARY:
Lichen planus is a chronic inflammatory mucocutaneous disease, which often results in oral manifestations, receiving the name of oral lichen planus (OLP). Its frequency varies from 0,1 to 4% of the general population, with a higher incidence in women, around the 4th and 5th decades of life. Although the pathogenesis of OLP is related to a immune-cellular response, mainly mediated by T lymphocytes, its cause remains unknown. Considering its chronic nature, control of OLP aims to reduce symptoms and improve function, and agents with anti-inflammatory action, especially topical corticosteroids result in some degree of success in most patients, depending on the clinical presentation. However, some cases are resistant to the use of corticosteroids, thus justifying the search for new therapeutic options. The immunomodulation proved to be one of the main functions of probiotic bacteria, and recent studies have shown effect of probiotics on decreasing the expression of inflammatory markers, which enables the study of this therapy as an alternative to the control of OLP. Thus, this project aims to evaluate the effects of therapy with Bifidobacterium animalis subsp. lactis HN019 comparing with clobetasol propionate 0.05% in symptomatic patients with OLP referred for diagnosis and treatment of School of Dentistry of Ribeirão Preto - University of São Paulo (USP). The impact of the topical therapy (probiotic or corticosteroid) on the clinical, histopathological and immunopathological features will be evaluated. This project was previously submitted and approved by the Institutional Review Board of the School of Dentistry of Ribeirão Preto/USP, and all patients must give informed consent to participate in this study.

DETAILED DESCRIPTION:
This is a randomized double-blind clinical trial with symptomatic patients presenting OLP, which will be randomly assigned to either topical Bifidobacterium animalis subsp lactis HN019 or clobetasol propionate 0.05%. The selected patients will receive capsules to be diluted in 15 ml of water containing 6 x 109 CFUs of Bifidobacterium subsp. lactis HN019 (experimental group) or 0.05% clobetasol propionate (control group) for mouth washing, twice a day for 4 weeks. Patients will be instructed to maintain normal brushing and not to use or consume another corticosteroid and /or probiotic during the study. Outcomes measures will be symptoms (VAS and Likert-like scale), quality of life (SF-36 form), and clinical changes (erythema, reticulation, erosion/ulcer based on clinical photographs), which will be performed at baseline, 15 days (only VAS, Likert-like scale and photographs) and and at one month of treatment. All patients will undergo biopsies for the diagnosis of OLP, and those who consent will be submitted to an optional biopsy at the end of the topical treatment for histopathological and immunopathological characterization.

ELIGIBILITY:
Inclusion Criteria:

* Clinical inclusion

  * Adults ≥ 18 years old, both genres, who consent to participate of the study;
  * Presence of symptomatic reticular lesion and/or white-gray papules. In afro-descendent individuals, reticular lesions may be associated with hyperpigmented lesions;
  * Additional clinical features such as ulcerative, erythematous, plaque and bullous lesions will be accepted in the presence of bilateral and symmetrical reticular lesions.
* Histopathological inclusion criteria

  * Presence of subepithelial infiltrate predominantly lymphocytic, in band and confined to the subepithelial area.
  * Liquefaction degeneration of the basal cells layer.

Exclusion Criteria:

* Clinical exclusion criteria

  * Exclusion of contact lichenoid lesions: the pattern of reticular lesion and / or papules should not be present only in areas of physical contact with restorative materials;
  * Exclusion of lichenoid reaction to the drug: difficult to differentiate from OLP, however it is necessary to report all drugs in use by the patient; the comparison between patients on medication, and those who do not use medication is important to establish subgroups of OLP;
  * Exclusion of chronic graft versus host disease (GVHD): differentiation between OLP and GVHD is established in most cases by medical history;
  * Exclusion of immunocompromised patients or patients with systemic diseases of high complexity.
  * Exclusion of patients who have previously used probiotic bacteria in the last 4 weeks prior to the study.
* Histopathological criteria for exclusion • Presence of epithelial dysplasia, absence of the lymphocytic inflammatory infiltrate band and liquefaction degeneration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2018-04-05 (Actual); Study Completion 2019-12-06 (Actual)

PRIMARY OUTCOMES:
Change in symptoms intensity measure | 4 weeks
  Self reported symptoms at baseline, 15 and 30 days after therapy through an visual analogue scale (VAS). It consists of a subjective scale scoring the symptoms from 0 to 10 (0 = no symptoms and 10 = as bad as can be).

SECONDARY OUTCOMES:
Histopathological analysis | Before (baseline) and one month after intensive topical therapy
  Biopsies will be collected at the baseline stage or at the time of the diagnosis of OLP (optional), consisting of a 5mm x 5mm fragment or a 4mm punch of reticular lesions. The second biopsy will be optional, with patient consent, close to the area of the first biopsy for comparative purposes. The histological findings will be determined quantitatively and qualitatively regarding the presence of epithelial hyperplasia, degeneration by liquefaction of the basal cells layer, lymphocytic infiltrate in the subepithelial connective tissue, and apoptotic cells. Photographs will be used at 400x and quantification using the Image J. program.
Immunohistochemical analysis | After 4 weeks of intensive therapy.
  The population of inflammatory cells will be characterized by analysis of oral mucosa samples, with emphasis on the T cell line (CD3, CD4, CD8, CD25, CD103, perforin, granzyme B and Foxp3), B cells (CD20 / CD20), dendritic cells (CD123 and CD303), submucosal dendritic cells (CD209 and factor XIIIa), Langerhans cells (CD1a and CD207), endothelial activity (e-selectin and CD31), mast cells ), macrophages (CD68 and CD163), myeloid dendritic cells (S100 and CD11c), cell proliferation markers (Ki-67, MCM-2, MCM-5, cyclin D1) and extracellular matrix (laminin-5). For immunohistochemical reactions, histological sections of 3μm thickness will be performed, which will be placed on slides coated with organosilane (Sigma-Aldrich, St Louis, MO, USA).
Venous blood collection | Before (baseline) and after 4 weeks of topical therapy
  10 ml of venous blood to evaluate the probiotic systemic effect, by means of the research of pro-inflammatory, anti-inflammatory and regulatory cytokines.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Reis Messora, DDS, PhD, Study Chair — University of São Paulo, Ribeirão Preto, SP, Brazil.; Sergio L. Souza Salvador, DDS, PhD, Study Chair — University of São Paulo, Ribeirão Preto, SP, Brazil.; Átila V. Vitor Nobre, DDS, Study Chair — University of São Paulo, Ribeirão Preto, SP, Brazil.; Cristhiam de J. Hernández Martínez, DDS, Study Chair — University of São Paulo, Ribeirão Preto, SP, Brazil.; Kleber Tanaka Suzuki, DDS, Study Chair — University of São Paulo, Ribeirão Preto, SP, Brazil.; Marina C. Gabriel Del Arco, Study Chair — University of São Paulo, Ribeirão Preto, SP, Brazil.; Lara Maria A Innocentini, DDS,PhD, Study Chair — University of São Paulo, Ribeirão Preto, SP, Brazil.; Gilberto A Silva, MS, Study Chair — University of São Paulo, Ribeirão Preto, SP, Brazil.; Ellen E Monteiro, Student, Study Chair — University of São Paulo, Ribeirão Preto, SP, Brazil
Locations (1):
- School of Dentistry of Ribeirão Preto, University of São Paulo, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Han X, Zhang J, Tan Y, Zhou G. Probiotics: A non-conventional therapy for oral lichen planus. Arch Oral Biol. 2017 Sep;81:90-96. doi: 10.1016/j.archoralbio.2017.04.026. Epub 2017 Apr 26. PMID 28499235
- [Background] Garcia-Pola MJ, Gonzalez-Alvarez L, Garcia-Martin JM. Treatment of oral lichen planus. Systematic review and therapeutic guide. Med Clin (Barc). 2017 Oct 23;149(8):351-362. doi: 10.1016/j.medcli.2017.06.024. Epub 2017 Jul 28. English, Spanish. PMID 28756997
- [Background] Sivaraman S, Santham K, Nelson A, Laliytha B, Azhalvel P, Deepak JH. A randomized triple-blind clinical trial to compare the effectiveness of topical triamcinolone acetonate (0.1%), clobetasol propionate (0.05%), and tacrolimus orabase (0.03%) in the management of oral lichen planus. J Pharm Bioallied Sci. 2016 Oct;8(Suppl 1):S86-S89. doi: 10.4103/0975-7406.191976. PMID 27829754
- [Background] Ricoldi MST, Furlaneto FAC, Oliveira LFF, Teixeira GC, Pischiotini JP, Moreira ALG, Ervolino E, de Oliveira MN, Bogsan CSB, Salvador SL, Messora MR. Effects of the probiotic Bifidobacterium animalis subsp. lactis on the non-surgical treatment of periodontitis. A histomorphometric, microtomographic and immunohistochemical study in rats. PLoS One. 2017 Jun 29;12(6):e0179946. doi: 10.1371/journal.pone.0179946. eCollection 2017. PMID 28662142
- [Background] Gerhard D, Sousa FJDSS, Andraus RAC, Pardo PE, Nai GA, Neto HB, Messora MR, Maia LP. Probiotic therapy reduces inflammation and improves intestinal morphology in rats with induced oral mucositis. Braz Oral Res. 2017 Jul 3;31:e71. doi: 10.1590/1807-3107BOR-2017.vol31.0071. PMID 28678976